CLINICAL TRIAL: NCT02778373
Title: Comparative Effects of Post-exercise Ingestion of a High or Low Molecular Weight Solution on Resistance Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 1401-45-1401
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Task Performance and Analysis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Flavored Water
  Interventions: Other: Placebo: Water
- Low Molecular Weight Carbohydrate (Active Comparator): low molecular weight carbohydrate delivered post-endurance exercise in a 10% solution providing 1.2 grams/kg body weight carbohydrate
  Interventions: Dietary Supplement: DE15 maltodextrin, Matrin® M160, Grain Processing Corporation, Muscatine, IA
- High molecular weight carbohydrate (Experimental): high molecular weight carbohydrate delivered post-endurance exercise in a 10% solution providing 1.2 grams/kg body weight carbohydrate
  Interventions: Dietary Supplement: Vitargo ®, Swecarb AB, Karlskrona, Sweden

INTERVENTIONS:
Dietary Supplement: Vitargo ®, Swecarb AB, Karlskrona, Sweden
  Arms: High molecular weight carbohydrate
Dietary Supplement: DE15 maltodextrin, Matrin® M160, Grain Processing Corporation, Muscatine, IA
  Arms: Low Molecular Weight Carbohydrate
Other: Placebo: Water
  Arms: Placebo

SUMMARY:
This study sought to examine differences in resistance exercise performance, as measured by the kinetic and kinematic profile during multiple sets of the back squat exercise, following ingestion of high or low molecular weight carbohydrate beverages.

ELIGIBILITY:
Inclusion Criteria:

* having at least 2 years resistance training experience to include the parallel back squat exercise at least once a week
* no musculoskeletal injury within previous 1 year
* not having consumed any nutritional or ergogenic supplement excluding protein and/or a daily vitamin for the previous 6-week period

Exclusion Criteria:

* no previous resistance training experience
* musculoskeletal injury within the previous 1 year
* having consumed or presenting consuming a nutritional or ergogenic supplement

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Power Output | 1 year
  Change in power output, measured in watts, will be examined over the course of the performance of 5 sets of 10 repetitions of the back squat exercise with a weight corresponding to 75% one-repetition maximum.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Piehl Aulin K, Soderlund K, Hultman E. Muscle glycogen resynthesis rate in humans after supplementation of drinks containing carbohydrates with low and high molecular masses. Eur J Appl Physiol. 2000 Mar;81(4):346-51. doi: 10.1007/s004210050053. PMID 10664095
- [Background] Leiper JB, Aulin KP, Soderlund K. Improved gastric emptying rate in humans of a unique glucose polymer with gel-forming properties. Scand J Gastroenterol. 2000 Nov;35(11):1143-9. doi: 10.1080/003655200750056600. PMID 11145284
- [Background] Stephens FB, Roig M, Armstrong G, Greenhaff PL. Post-exercise ingestion of a unique, high molecular weight glucose polymer solution improves performance during a subsequent bout of cycling exercise. J Sports Sci. 2008 Jan 15;26(2):149-54. doi: 10.1080/02640410701361548. PMID 17852670
- [Derived] Oliver JM, Almada AL, Van Eck LE, Shah M, Mitchell JB, Jones MT, Jagim AR, Rowlands DS. Ingestion of High Molecular Weight Carbohydrate Enhances Subsequent Repeated Maximal Power: A Randomized Controlled Trial. PLoS One. 2016 Sep 16;11(9):e0163009. doi: 10.1371/journal.pone.0163009. eCollection 2016. PMID 27636206